CLINICAL TRIAL: NCT02980640
Title: Swiss Multiple Sclerosis Registry
Acronym: SMSR
Status: Recruiting | Type: Observational
Sponsor: Swiss Multiple Sclerosis Registry (Other)
Collaborators: University of Zurich (Other); Schweizerische Multiple Sklerose Gesellschaft (Other)
Responsible Party: Sponsor
Other Study IDs: PB_2016-00894
Record Dates: First submitted 2016-11-23; First posted 2016-12-02 (Estimated); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis; Treatment; Quality of Life; Symptoms
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 25 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The Swiss Multiple Sclerosis Registry is a national, patient-centered registry with the aim to document the epidemiology of multiple sclerosis (MS), as well as the quality of life of persons living with MS in Switzerland.

DETAILED DESCRIPTION:
The Swiss Multiple Sclerosis Registry is a national, patient-centered research project with the aim to document the epidemiology of multiple sclerosis (MS), as well as the quality of life of persons living with MS in Switzerland. The Swiss MS Registry pursues a "Citizen Science" approach, that is, persons with MS are not just study participants but also act as MS experts and are active contributors to the interdisciplinary Swiss MS Registry research network. Initiated and funded by the Swiss MS Society, the Swiss MS Registry represents a collaborative effort by numerous MS caregivers, researchers and persons with MS. It is hosted by the Epidemiology, Biostatistics and Prevention Institute at the University of Zurich.

How many MS-affected persons are living in Switzerland and how are they coping with MS in their daily lives? What is the current situation with regard to access to and use of drug and non-drug treatments for MS? These and other questions are addressed by means of semi-annual surveys. Further research activities concern the quality of life of persons with MS, mobility, personal resources and support by friends and family, work situation, mental health, clinical progression of MS, as well as alternative therapies.

Owing to a flexible study design, participants can decide between different levels of commitment (from one-time surveys to repeated, semiannual surveys and medical records review). Furthermore, study participants receive summaries of their data as charts and tables. Data collection primarily occurs via a newly designed online platform, but paper-and-pencil questionnaires are also available. As an additional incentive, the online platform includes a diary with basic capabilities for analyses and printing.

ELIGIBILITY:
Inclusion Criteria:

* Persons with a confirmed Multiple Sclerosis Diagnosis
* 18 years and older
* Living in Switzerland or receiving MS care in Switzerland

Exclusion Criteria:

* Younger than 18 years
* Not living in Switzerland and not receiving MS care in Switzerland

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All persons with Multiple Sclerosis who either live in Switzerland or who recieve MS care in Switzerland
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2016-06; Primary Completion 2041-06 (Estimated); Study Completion 2041-06 (Estimated)

PRIMARY OUTCOMES:
Change in Health-Related Quality of Life | Baseline; 6, 12, 18, 24, 30, 36, 42, 48, 54, 60 months
  Assessment via EQ-5D
Change in Self-Assessment of Health Status | Baseline; 6, 12, 18, 24, 30, 36, 42, 48, 54, 60 months
  Assessment via Visual Analogue Scale

SECONDARY OUTCOMES:
Occurrence of MS Symptoms | Baseline; 6, 12, 18, 24, 30, 36, 42, 48, 54, 60 months
  Self-report of new and recurrent MS symptoms
Occurrence of Adverse Drug Effects | Baseline; 6, 12, 18, 24, 30, 36, 42, 48, 54, 60 months
  Self-report of unwanted drug side effects
Occurrence of MS Relapse | Baseline; 6, 12, 18, 24, 30, 36, 42, 48, 54, 60 months
  Self-report of MS relapse(s)

CONTACTS AND LOCATIONS:
Overall Officials: Milo Puhan, MD PhD, Principal Investigator — University of Zurich
Locations (1):
- University of Zurich; Epidemiology, Biostatistics & Prevention Institute, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
Pseudonimized data are shared with other researchers upon approval of a project proposal. Guidelines describing submission and approval process are in place.

REFERENCES:
- [Derived] Kamm CP, Barin L, Gobbi C, Pot C, Calabrese P, Salmen A, Achtnichts L, Kesselring J, Puhan MA, von Wyl V; Swiss Multiple Sclerosis Registry (SMSR). Factors influencing patient satisfaction with the first diagnostic consultation in multiple sclerosis: a Swiss Multiple Sclerosis Registry (SMSR) study. J Neurol. 2020 Jan;267(1):153-161. doi: 10.1007/s00415-019-09563-y. Epub 2019 Oct 8. PMID 31595377
- [Derived] Steinemann N, Kuhle J, Calabrese P, Kesselring J, Disanto G, Merkler D, Pot C, Ajdacic-Gross V, Rodgers S, Puhan MA, von Wyl V; Swiss Multiple Sclerosis Registry. The Swiss Multiple Sclerosis Registry (SMSR): study protocol of a participatory, nationwide registry to promote epidemiological and patient-centered MS research. BMC Neurol. 2018 Aug 13;18(1):111. doi: 10.1186/s12883-018-1118-0. PMID 30103695
- See also: Description of Swiss MS Registry in German — http://www.ms-register.ch
- See also: Description of Swiss MS Registry in French — http://www.registre-sep.ch
- See also: Description of Swiss MS Registry in Italian — http://www.registro-sm.ch
- See also: Protocol Description of the Swiss Multiple Sclerosis Registry — https://bmcneurol.biomedcentral.com/articles/10.1186/s12883-018-1118-0